CLINICAL TRIAL: NCT00567463
Title: Early Anti-inflammatory Treatment of Asymptomatic or Mildly Symptomatic Airway Hyperresponsiveness
Brief Title: Early Antiinflammatory Treatment of Asthma
Acronym: EATA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Completed
Sponsor: Laval University (Other)
Responsible Party: Louis-Philippe Boulet, Laval Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HL-EATA-550
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2007-12

CONDITIONS: Asthma; Bronchial Hyperreactivity
Keywords: Asthma; Bronchial hyperresponsiveness; Methacholine; Induced sputum; bronchial biopsies
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (Placebo Comparator): Placebo inhalator will be used by subjects in the placebo group(same course as patients in the treated group)
  Interventions: Device: Fluticasone

INTERVENTIONS:
Device: Fluticasone — Fluticasone 250mcg for 3 months followed by 100mcg for 9 months, one puff once a day at supper time

SUMMARY:
* The inflammatory process that leads to the development of asthma may be present before the onset of asthma symptoms and cause a certain degree of airway hyperresponsiveness. Without treatment it may induce irreversible airway structural changes that are associated with permanent changes in airway functions, persistent airway hyperresponsiveness and lead to the development of asthma symptoms.
* Atopic subjects with asymptomatic airway hyperresponsiveness and first degree relatives with a history of asthma are at higher risk to develop symptomatic asthma. Early treatment of airway inflammation in these predisposed subjects with " borderline " or mild airway hyper-responsiveness could prevent the development of asthma symptoms, and reduce or even normalize airway responsiveness.
* In very mild asthmatic subjects (bronchodilator need < thrice a week), early anti-inflammatory treatment can lead to " normalisation " or airway responsiveness in a significant number of subjects and prevent the need for subsequent regular therapy. This is particularly true for those showing blood/sputum eosinophilia.

Objectives: To compare perception of bronchoconstriction, pulmonary function and airway inflammation in subjects with mild symptomatic asthma and asymptomatic asymptomatic airway hyperresponsiveness

Methods: To compare the influence of inhaled fluticasone propionate 250 mcg/day for 3 months followed by 100 mcg/day for 9 months on airway inflammation and methacholine responsiveness in a double-blind, placebo-controlled, parallel groups study including non-smoking atopic subjects with mild asthma and asymptomatic airway hyperresponsiveness

DETAILED DESCRIPTION:
* Evaluate the change in airway hyperresponsiveness and in inflammatory markers in the blood and sputum in the population studied following a 3-month course of fluticasone 250 µg per day followed by a 9-month course of fluticasone 1000 µg per day (before supper) compared to placebo as measured on a regular basis over a two year period.
* This study will include:

  1. A baseline evaluation period of 2 weeks before starting the 3-month treatment period followed by the 9-month treatment period.
  2. Treatment will be double-blinded, randomized, parallel design.
  3. A follow-up period of one year.

Optional: Bronchoscopies with bronchial biopsy sampling will be performed before and after tratment in a subgroup of subjects to determine what is the influence of this corticosteroid treatment on airway inflammation and remodelling.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 to 45 years old.
2. Methacholine PC20 0,5-16 mg/ml and FEV1 greater than 80% pred.
3. Asymptomatic AHR patients will have had no past or present symptoms of intermittent dyspnea or wheezing, chronic cough or phlegm production as defined by negative responses to the European community respiratory health survey (ECRHS) questionnaire. They will also never have experienced symptoms similar to those induced by the methacholine challenge (misinterpretation of asthma symptoms).

   Subjects with mild intermittent symptoms will have had asthma symptoms less than twice a week in the last 3 months. They will, however, demonstrate variable airflow obstruction according to the Canadian asthma consensus criteria. They will have required asthma medication at least occasionnally within the last year.
4. At least one positive response to indoor allergens (cats, dogs, housedust mites or cockroach).
5. At least one first degree relative with asthma.
6. Current exposure to a dog or a cat at home.
7. FEV1 greater than 80% of predicted (Knudson 1983).

Exclusion Criteria:

1. Subjects who have used inhaled corticosteroids or any other bronchial anti-inflammatory agents in the past.
2. Subjects who smoked more than 6 packs/year, or who smoked in the last twelve months.
3. Poor-perceivers of airflow obstruction (Borg score = 1 on methacholine challenge at 20% fall in FEV1).
4. Women either pregnant or breastfeeding or those without adequate contraception.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 1998-12; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in airway hyperresponsiveness in the population studied following 3-month of fluticasone 250 µg per day followed by 9-month of fluticasone 1000 µg per day compared to placebo. | measurements every 3 months for 2 years

SECONDARY OUTCOMES:
- Evaluate the change in inflammatory markers in blood and sputum vs placebo. - Determine if this treatment will reduce asthma symptoms over a period of 2 years. - Determine its influence on airway inflammation and remodelling (bronchial biopsies). | measurements every 3 months during two years

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Hôpital Laval
Locations (1):
- Centre de Recherche, Hôpital Laval, Québec, Quebec, Canada